CLINICAL TRIAL: NCT01350232
Title: Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation for Sickle Cell Anemia From HLA Matched or Partially-Matched Related Donors
Brief Title: Treatment of Sickle Cell Anemia With Stem Cell Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09F.327; 1-RC2HL101496-0 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute); JT 1526 (Other: JeffTrial Number); 1RC2HL101496 (NIH)
Record Dates: First submitted 2011-05-04; First posted 2011-05-09 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Anemia; Sickle Cell-hemoglobin C Disease; Sickle Cell-β0-thalassemia
Keywords: sickle cell; SS disease; SC disease; S-thalassemia; transplant; bone marrow transplant; stem cell transplant; matched sibling; haploidentical; hemoglobinopathy; anemia; desensitization
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease; Hemoglobinopathies; Anemia | interventions — fludarabine; fludarabine phosphate; Cytarabine; Whole-Body Irradiation; Cyclophosphamide; Bortezomib; Rituximab; Plasmapheresis; Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HSCT (Experimental): Subjects receive the preparative regimen in 2 steps. The "first step" will be with fludarabine and cytarabine and a low dose of total body irradiation. This will be followed by the "first step" of the transplant graft - the donor lymphocytes. The "second step" of the chemotherapy will be two doses of cyclophosphamide. This will then be followed by the "second step" of the transplant graft - the stem cells.
  Only subjects with prior alloimmunization against donor will receive desensitization. Subjects who demonstrate alloimmunization against the HLA of the donor will receive bortezomib and rituximab in combination with plasmapheresis prior to the admission for transplant.
  Interventions: Drug: Fludarabine; Drug: Cytarabine; Device: Cellular Infusions; Radiation: Total Body Irradiation; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Rituximab; Procedure: Plasmapheresis

INTERVENTIONS:
Drug: Fludarabine — Subjects will receive fludarabine at a dose of 30 mg/m2 daily for 4 days as part of the preparative regimen
  Other Names: Fludara
Drug: Cytarabine — Subjects will receive cytarabine at a dose of 2 g/m2 daily for 4 days, approximately 4 hours after the fludarabine
  Other Names: Ara-C; Cytosar; Cytosine arabinoside
Device: Cellular Infusions — Subjects will receive the cellular product in 2 steps. The first is a lymphocyte infusion of 2 X 10e8 lymphocytes/kg on the day they receive total body irradiation. The second is a CD34 enriched stem cell product approximately 48 hours after the cyclophosphamide.
  The CliniMACS® Plus Instrument will be used for the selection of human CD34+ hematopoietic stem and progenitor cells in human allogeneic hematopoietic stem cell transplantation.
  Other Names: Stem Cells; DLI; HPCT
Radiation: Total Body Irradiation — All subjects will receive 200cGy TBI in a single fraction on the AM they receive the lymphocyte infusion
  Other Names: TBI
Drug: Cyclophosphamide — All subjects will receive cyclophosphamide at a dose of 60 mg/kg at approximately 72 and 96 hours after the lymphocyte infusion
  Other Names: Cytoxan
Drug: Bortezomib — Subjects will receive bortezomib 1.3 mg/kg on Day 1,4,8, and 11 of a 21 day cycle. This will be repeated for 2 cycles.
  Other Names: Velcade
Drug: Rituximab — Subjects will receive rituximab 375 mg/m2 on day 1 and day 8 of a 21 day cycle, on days they will also be receiving rituximab. This will be repeated for 2 cycles.
  Other Names: Rituxan
Procedure: Plasmapheresis — Subjects who continue to have detectable anti-donor antibody will receive plasmapheresis to reduce the antibody further
  Other Names: Plasma exchange

SUMMARY:
This is a clinical research trial in which a novel preparatory regimen was developed for bone marrow transplant (BMT) which eliminates the primary obstacle to transplant, the lack of a matched sibling donor. It is believed this regimen is sufficiently efficacious and sufficiently gentle to apply to patients with sickle cell anemia and related disorders. It is proposed to characterize the efficacy and toxicity of this regimen in high risk patients with sickle cell anemia using criteria for patient selection that have been accepted in prior BMT trials in patients with sickle cell disease, specifically only the subset of patients whose prior clinical behavior indicates that they are at high risk for serious morbidity and early mortality. In addition, it is proposed to characterize the pathophysiology of a consistent febrile response seen in the haploidentical BMT regimen the investigators have developed at Thomas Jefferson University (TJU).

The primary goal of this study is to determine the response rate to a reduced intensity conditioning regimen which consists of fludarabine, cytarabine, low dose total body irradiation and cyclophosphamide in patients with severe sickle cell anemia.

DETAILED DESCRIPTION:
Hemoglobinopathies, such as sickle cell disease and thalassemia major, constitute a group of genetic diseases associated with significant morbidity and premature death. In the 1970s, the mean survival of patients with sickle cell disease was 14.3 years. With improvements in medical practice, this has improved such that estimates are now into the third decade of life.

In patients with sickle cell disease, a single amino acid substitution in beta-hemoglobin causes erythrocytes to sickle in response to oxidative stress. The sequelae of this defect are vaso-occlusive crises, resulting in episodes of bony pain and infarction, acute chest syndrome, and strokes. Life long need for transfusion leads to complications including alloimmunization and iron overload. The latter condition is frequently associated with significant end-organ damage.

In recent years, new strategies in supportive care, such as the use of hydroxyurea to stimulate fetal hemoglobin production in patients with sickle cell anemia, have resulted in the amelioration of some of the devastating manifestations of this disease. However, this therapy does not benefit all patients, and there have been concerns about the possible risk of latent transformation to leukemia with prolonged use of this drug. Clearly, better treatment strategies are needed for this devastating group of diseases.

Patients with sickle cell anemia will be offered enrollment on a clinical trial of reduced intensity stem cell transplant. The transplant donors will be either HLA matched siblings or family members who are 50% matched for HLA. Patients will receive therapy in 2 steps.

For patients who are allo-immunized against the donor (patients who have made an immune response already against the donor's HLA type), there will be a desensitization process. This will be outpatient therapy and will include therapy with bortezomib on the 1st, 4th, 8th and 11th day of a 21 day cycle. This will be repeated for a second cycle, for a total of 8 doses of bortezomib over a 6 week period. In addition, they will receive rituximab on the 1st and 8th day of each cycle. These therapies are designed to decrease the subject's chance of rejecting the transplant, as it is known that patients with sickle cell anemia are likely to be heavily immunized against donors. For patients who have high levels of antibodies against the donors, a plasmapheresis procedure will be performed prior to admission as well. All patients will undergo red cell exchange prior to admission.

During the transplant admission, subjects will receive a "Two Step" chemotherapy and transplant regimen. The chemotherapy "first step" will be with fludarabine and cytarabine and a low dose of total body irradiation. This will be followed by the "first step" of the transplant graft - the donor lymphocytes. The "second step" of the chemotherapy will be two doses of cyclophosphamide. This will then be followed by the "second step" of the transplant graft - the stem cells.

ELIGIBILITY:
Inclusion Criteria:

Patient Selection:

i) Patients with sickle cell disease (sickle cell anemia, sickle cell-hemoglobin C disease, or sickle cell-β0-thalassemia) confirmed by hemoglobin electrophoresis.

ii) Patients should have one or more of the following:

1. History of acute chest syndrome requiring recurrent hospitalization or exchange transfusion (Acute chest syndrome is defined as pulmonary infiltrate involving at least one complete lung segment, consistent with alveolar consolidation but not atelectasis, accompanied by chest pain, fever, cough, tachypnea or wheezing)
2. History of nonhemorrhagic stroke or central nervous system event lasting longer than 24 hours
3. Recurrent vaso-occlusive pain (≥5 episodes during the past two years) or recurrent priapism requiring hospitalization or visits to the emergency room or sickle cell day unit
4. Sickle nephropathy (moderate or severe proteinuria or a glomerular filtration rate 30-50% of normal predicted value) with progression on ACE inhibitor therapy iii) Patient must have failed therapy with hydroxyurea, as HU as evidenced by at least 6 months of maximum HU dosage for sickle cell disease, i.e. dose escalation to a level which caused some minimal hematologic toxicity in terms of CBC values. Failure to respond must also be documented by no significant increase in subjects HbF levels at this maximally tolerated dosage.AND development/ persistence of items listed in (ii) Patients who are deemed not eligible for hydroxyurea by the primary hematologist will be considered eligible without having failed hydroxyurea. Non-eligibility for hydroxyurea therapy is based on:

(1) the diagnoses of SC disease and sickle cell-β0-thalassemia in which no clear evidence supports the use of hydroxyurea therapy and thus treatment with hydroxyurea is not considered the standard of care in these entities (2) the presence of high hemoglobin F levels in patients with sickle cell anemia and documented Hereditary Persistence of Fetal Hemoglobin (HPFH) in which hydroxyurea is not considered the standard of care (3) severe adverse reactions to hydroxyurea in patients with sickle cell anemia based on, but not limited to, count suppression, GI intolerance, and dermatomyositis Patient unwillingness to be compliant with hydroxyurea therapy is not an acceptable reason for non-eligibility iv) Patients must have an acceptable related donor

1. who is matched at the HLA-A;B; C; DR loci (8 of 8 match) or mismatched for at most one locus (7 of 8 match) (well matched related donor
2. who is mismatched at 2-4 alleles (haplo-identical) v) Patient age greater than 18 - 45 years vi) ECOG performance status 0-2/ Karnofsky 70-100% vii) Written informed consent obtained from the patient. viii) Transaminases <3X ULN; patients with transaminases greater than the ULN but less than 3XULN will be evaluated by the hepatology service and will undergo further imaging and biopsy as deemed necessary by hepatology. They will not be considered eligible unless cleared by hepatology.

Exclusion Criteria:

Patient Selection:

i) Pregnancy/ unwillingness to use adequate contraception during study period ii) Liver disease including

1. Acute hepatitis (transaminases >3x normal value)
2. Chronic hepatitis C
3. Chronic hepatitis B or history of exposure to hepatitis B iii) Cardiac ejection fraction < 50% iv) Pulmonary hypertension - as evidenced by findings on resting echocardiogram of pulmonary artery systolic pressure ≥ 40 mmHg or any evidence of right ventricular dysfunction (hypokinesis or RV dilation) v) Severe renal impairment (GFR <30% of predicted normal value) vi) Severe residual functional neurologic impairment (other than hemiplegia alone) vii) DLCO ≤50 viii) Any evidence of infection by the human immunodeficiency virus ix) Psychiatric disorder that would preclude patients from signing an informed consent x) Severe neuro-cognitive or executive function making informed consent possible

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Filicko-O'Hara, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org

RESULTS

PARTICIPANT FLOW:
Groups:
- HSCT: Subjects receive the preparative regimen in 2 steps. The "first step" will be with fludarabine and cytarabine and a low dose of total body irradiation. This will be followed by the "first step" of the transplant graft - the donor lymphocytes. The "second step" of the chemotherapy will be two doses of cyclophosphamide. This will then be followed by the "second step" of the transplant graft - the stem cells.
  Only subjects with prior alloimmunization against donor will receive desensitization. Subjects who demonstrate alloimmunization against the HLA of the donor will receive bortezomib and rituximab in combination with plasmapheresis prior to the admission for transplant.
  Fludarabine: Subjects will receive fludarabine at a dose of 30 mg/m2 daily for 4 days as part of the preparative regimen
  Cytarabine: Subjects will receive cytarabine at a dose of 2 g/m2 daily for 4 days, approximately 4 hours after the fludarabine
  Cellular Infusions: Subjects will receive the cellular
Period: Overall Study
Arm/Group | HSCT
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HSCT
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (3.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Stable Engraftment
Description: To determine if the reduced intensity preparative regimen of fludarabine, cytarabine, cyclophosphamide and low-dose total body irradiation will generate stable engraftment with donor hematopoietic stem cells in at least 80% of patients with severe sickle cell anemia.
Time Frame: 180 days post-infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

2. Secondary Outcome: Organ Toxicity
Description: To assess organ toxicity related to fludarabine, cytarabine, cyclophosphamide and low-dose total body irradiation in a population with severe sickle cell anemia.
Time Frame: 30 days post infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: To determine the overall survival at 6 months post-transplant in patients receiving a matched or partially-matched related donor transplant after reduced-intensity conditioning.
Time Frame: 6 months post infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

4. Secondary Outcome: Acute Graft Versus Host Disease
Description: To describe the incidence and severity of acute and chronic GVHD following this reduced intensity transplant from partially matched related donors using a combination of cyclophosphamide, tacrolimus and mycophenolate mofetil (MMF) as GVHD prophylaxis.
Time Frame: 100 days post infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

5. Secondary Outcome: Correction of Hemoglobinopathy
Description: To evaluate the extent of correction of hemoglobinopathy following this reduced intensity transplant.
Time Frame: 100 days post infusion through 5 years post infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

6. Secondary Outcome: Immune Recovery
Description: To assess the pace of lymphoid recovery and associated risk for opportunistic infections and relapse (return to recipient erythropoiesis) in this patient population.
Time Frame: 100 days post infusion through 5 years post infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

7. Secondary Outcome: Quality of Life
Description: To describe the quality of life and functional status following transplantation.
Time Frame: Through 5 years post infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

8. Secondary Outcome: Cytokine Profile
Description: To characterize the profiles of cytokines released following administration of the lymphoid portion of the transplant (donor lymphocyte infusion [DLI]).
Time Frame: Through 5 years after infusion
Arm/Group | HSCT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | HSCT
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSCT (N=2)
Chest pain (General disorders) | 1 (1)
Knee pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HSCT (N=2)
Abdominal cramps (General disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Back pain (General disorders) | 1 (1)
Bone pain (General disorders) | 1 (1)
CMV reactivation (Immune system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Migraine (General disorders) | 1 (1)
Nausea (General disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Tingling in fingers/toes (General disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to poor accrual. No reportable data has been collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes